CLINICAL TRIAL: NCT05211193
Title: Open Label, Multi Center Study to Evaluate the Efficacy of the Home Based Electrical Transcutaneous NeuroModulation (eTNM) Treatment Via Nerve Stimulator URIS I (Tesla Medical) in the Treatment of Overactive Bladder (OAB).
Brief Title: Open Label Study to Evaluate the Efficacy of the Home Based Electrical Transcutaneous URIS I in the Treatment of Overactive Bladder (OAB).
Status: Completed | Type: Observational
Sponsor: Stimvia s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: TS003
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Overactive Bladder (OAB); Failed Any OAB Pharmacotherapy
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- eTNM arm: eTNM delivered by URIS I nerve stimulation device, self administered in the subject's home for 30 minutes per day, for a minimum of 34 therapy session between day 1- 42.
  Interventions: Device: eTNM delivered by URIS I nerve stimulation device

INTERVENTIONS:
Device: eTNM delivered by URIS I nerve stimulation device — eTNM delivered by URIS I nerve stimulation device, self administered in the subject's home for 30 minutes per day, for a minimum of 34 therapy session between day 1-42.

SUMMARY:
Open label Study to Evaluate the Efficacy of the Home Based Electrical Transcutaneous NeuroModulation (eTNM) Treatment Via Nerve Stimulator URIS I in the Treatment of Overactive Bladder.

DETAILED DESCRIPTION:
Open label, Multi center Study to Evaluate the Efficacy of the Home Based Electrical Transcutaneous NeuroModulation (eTNM) Treatment Via Nerve Stimulator URIS I in the Treatment of Overactive Bladder (OAB).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older, inclusive
* Diagnosis of OAB or mixed incontinence with the predominance of OAB symptoms
* Dissatisfaction with any current or previous pharmacotherapy treatment of OAB for any reason within the past 12 months
* Treatment Satisfaction VAS <50
* Ability to understand and sign ICF
* Subject agreed to attend all follow up evaluations and was willing to completely and accurately fill out voiding diaries and questionnaires, and was willing to complete required exams and tests
* Subject agreed not to participate in another research study from the time of screening until the final study visit
* Subject agreed not to use a pharmacotherapy treatment for OAB from the time of screening until the final study visit

Exclusion Criteria:

* Prior treatment with botulotoxin for OAB
* Previous pharmacotherapy for OAB if >12 months ago
* Urinary retention with post void residual > 150ml
* Neurological disease affecting urinary bladder function, including but not limited to Parkinson's disease, multiple sclerosis, stroke, spinal cord injury and nerves of lower limbs
* History or presence of stress incontinence, or mixed incontinence where stress incontinence was predominant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: females age 18 years or older. The women had a diagnosis of OAB or mixed incontinence with the predominance of OAB symptoms. The women were dissatisfied with current or previous pharmacotherapy treatment of OAB for any reason within the past 12 months.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Change of severe urgency episodes | baseline and end of study (6weeks treatment)
  The proportion of subjects with ≥ 50% change in severe urgency episodes (Grade 3 or 4) will be summarized by visit and for the full treatment period using the last observation.

CONTACTS AND LOCATIONS:
Locations (1):
- MUDr. Michal Rejchrt, Příbram, Czech, Czechia

IPD SHARING:
Plan to Share IPD: No